CLINICAL TRIAL: NCT01934309
Title: Does Providing Medical Personnel in the AMPATH Network With Patient-specific Reminders Regarding TB That Are Generated From a Patient's EMR Improve the Prevalence of IPT Initiation and Decrease the Time From Screening to Treatment?
Brief Title: Clinical Decision-support Reminders to Improve IPT Initiation Among HIV Positive Adults in Western Kenya
Acronym: TBTech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Moi University (Other); Academic Model Providing Access to Healthcare (AMPATH) (Other); Regenstrief Institute, Inc. (Other); Innovative Support to Emergencies, Diseases and Disasters (InSTEDD) (Unknown); Kijani Consulting (Unknown)
Responsible Party: Principal Investigator, Paul Biondich, Associate Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: AID-OAA-TO-11-00060
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Tuberculosis
Keywords: tuberculosis; isoniazid preventative therapy; clinical decision support; HIV; Kenya; eHealth
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TB reminders (Experimental): Receive existing reminders plus new patient-specific reminders about TB screening, prevention, and treatment
  Interventions: Behavioral: TB reminders
- No TB reminders (No Intervention): Only receive existing reminders; no TB reminders

INTERVENTIONS:
Behavioral: TB reminders — The intervention to be studied involves providing clinic-based medical care providers (e.g., nurses, clinical officers, medical officers, consultants) with patient-speciﬁc clinical reminders regarding TB that are generated from a patient's electronic medical record and based on accepted clinical algorithms for TB screening and treatment.
  Arms: TB reminders

SUMMARY:
The overall research objective is to evaluate the impact of implementing a reminder system for medical providers to improve TB case-finding and isoniazid preventative therapy (IPT) for adults living with HIV in western Kenya

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the impact of implementing a clinical decision support reminder system for medical providers (i.e., nurses, clinical officers, medical officers, consultants) to improve tuberculosis case-ﬁnding and the use of isoniazid preventative therapy for adults living with HIV in western Kenya.

ELIGIBILITY:
Clusters:

Inclusion Criteria

* active
* uses HIV initial and return encounter paper forms
* enters data into the AMPATH medical records system (AMRS) or sends forms to central location for data entry
* prints or receives printed paper summary sheets with reminders
* interprets chest x-rays
* interprets sputum smear results
* prescribes IPT and dispenses INH
* completed an average of 10 initial adult HIV positive encounters per month in 2012
* HIV Care Clinic

Exclusion Criteria -

Patients:

Inclusion Criteria

* HIV positive
* complete an adult initial encounter at an HIV Care Clinic during the enrollment period
* attend at least one additional appointment within 90 days after the initial encounter

Exclusion Criteria

- history of TB or IPT

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3782 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Prescription of Isoniazid | within 3 months of initial encounter
  Provider prescribes INH within 3 months of patient's initial encounter.

SECONDARY OUTCOMES:
Time to isoniazid prophylactic therapy (IPT) initiation | within 3 months of initial encounter
  The time in weeks from a patient's initial encounter to the week the patient picks up the initial batch of INH from the pharmacy.

OTHER OUTCOMES:
Initiation of isoniazid prophylactic therapy (IPT) | within 3 months of initial encounter
  IPT will be considered "initiated" when a patient picks up the initial batch of the prescribed medications within 3 months of the initial encounter.
Isoniazid prophylactic therapy (IPT) completion | 9 months after treatment initiation
  Patient completes 9-month course of IPT

CONTACTS AND LOCATIONS:
Overall Officials: Lameck O Diero, MBChB, MMed, Principal Investigator — Moi University College of Health Sciences
Locations (1):
- AMPATH, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Green EP, Catalani C, Diero L, Carter EJ, Gardner A, Ndwiga C, Keny A, Owiti P, Israelski D, Biondich P. Do clinical decision-support reminders for medical providers improve isoniazid preventative therapy prescription rates among HIV-positive adults? Study protocol for a randomized controlled trial. Trials. 2015 Apr 9;16:141. doi: 10.1186/s13063-015-0558-8. PMID 25885266